CLINICAL TRIAL: NCT02145754
Title: Comparison of Two Culture Media for Cultivation of Borrelia Burgdorferi Sensu Lato
Brief Title: Culture Media for Borrelia Burgdorferi Sensu Lato
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana School of Medicine, Slovenia (Other)
Responsible Party: Principal Investigator, Franc Strle, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MKP,BSK-0613
Record Dates: First submitted 2013-06-24; First posted 2014-05-23 (Estimated); Results first posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Erythema Migrans
Keywords: erythema migrans; Lyme borreliosis; Borrelia burgdorferi; skin culture; culture media
MeSH Terms: conditions — Glossitis, Benign Migratory; Lyme Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MKP media versus BSK-H media (Active Comparator): one half of skin specimen obtained from erythema migrans patients was cultivated for Borrelia burgdorferi sensu lato in MKP media and the other half in BSK-H media
  Interventions: Other: MKP media; Other: BSK-H media

INTERVENTIONS:
Other: MKP media — one half of skin specimen was put in MKP media
Other: BSK-H media — one half of skin specimen was put in BSK-H media

SUMMARY:
The main purpose of this study is to compare effectiveness of two different culture media for cultivation of Borrelia burgdorferi sensu lato from skin specimens obtained from patients with erythema migrans.

ELIGIBILITY:
Inclusion Criteria:

* erythema migrans in patients > 18 years

Exclusion Criteria:

* pregnancy or lactation
* taking antibiotic with antiborrelial activity within 10 days
* erythema migrans localized on face or neck

Each patient (235 subjects) provided two skin samples (470 skin samples).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franc Strle, MD, PhD, Study Director — UMC Ljubljana; Eva Ruzic-Sabljic, MD, PhD, Principal Investigator — University of Ljubljana School of Medicine, Slovenia
Locations (1):
- UMC Ljubljana, Department of Infectious Diseases, Ljubljana, Slovenia

RESULTS

PARTICIPANT FLOW:
Groups:
- MKP Media Versus BSK-H Media: cultivation of Borrelia burgdorferi sensu lato (from skin specimens obtained from erythema migrans patients) in MKP media and in BSK-h media
  MKP media versus BSK-H media
Period: Overall Study
Arm/Group | MKP Media Versus BSK-H Media
Started | 235
Completed | 235
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MKP Media Versus BSK-H Media
Number analyzed (Participants) | 235
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 158
  >=65 years | 77
Age, Continuous [Mean (Full Range); unit: years] | 57 [21 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141
  Male | 94
Region of Enrollment [Number; unit: participants]
  Slovenia | 235

OUTCOME MEASURES:

1. Primary Outcome: Detection of Borrelia Burgdorferi Sensu Lato by Microscopy in Dark Field (Positive vs. Negative)
Description: number of erythema migrans skin samples with Borrelia Burgdorferi sensu lato detected by Microscopy in Dark Field
Time Frame: weekly examination during 9 weeks of cultivating for individual specimen
Population: Each participant provided two skin samples for analysis, one sample was cultivated in MKP, the other in BSK-H media.
Measure: Number; unit: culture-positive skin samples
Arm/Group | MKP Media Versus BSK-H Media
Number analyzed (Participants) | 235
culture-positive skin samples
  MKP media | 102
  BSK-H media | 59

ADVERSE EVENTS:
Arm/Group | MKP Media Versus BSK-h Media
Serious Adverse Events (participants affected / at risk) | 0/235
Other Adverse Events (participants affected / at risk) | 0/235

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes